CLINICAL TRIAL: NCT02034669
Title: A Phase II Study of Transplantation of Autologous Adipose Derived Stem Cells (ADSCs) in Completely Acute Spinal Cord Injury.
Brief Title: Transplantation of Autologous Adipose Derived Stem Cells (ADSCs) in Spinal Cord Injury Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri Phuoc Biotechnology., JSC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-VD-2012
Record Dates: First submitted 2014-01-06; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Acute Spinal Cord Injury
Keywords: Acute Spinal cord Injury, Adipose derived stem cells
MeSH Terms: interventions — Laminectomy; Injections, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with ADSCs transplantation (Experimental): 4 Intervention: laminectomy, intradural space at damage site, intrathecal at lumbar puncture, intravenous
  Interventions: Device: Laminectomy; Device: Intradural space; Device: Intrathecal; Device: Intravenous
- Treatment without ADSCs transplantation (No Intervention): Only intervention: laminectomy

INTERVENTIONS:
Device: Laminectomy — surgical laminectomy with glial scar resection
  Arms: Treatment with ADSCs transplantation
Device: Intradural space — ADSCs injection into Intradural space at damage site
  Arms: Treatment with ADSCs transplantation
Device: Intrathecal — ADSCs Intrathecal into lumbar puncture
  Arms: Treatment with ADSCs transplantation
Device: Intravenous — ADSCs intravenous
  Arms: Treatment with ADSCs transplantation

SUMMARY:
This study is designed to assess the safety and effect of autologous adipose derived stem cell (ADSCs) transplantation in acute spinal cord injury patients.

1. To assess the safety of autologous ADSCs transplantation in acute spinal cord injury and the complication after ADSCs transplantation.
2. To evaluate the effect of ADSCs isolation and expansion procedure.
3. To determine if functional outcome is improved following ADSCs transplantation in acute spinal cord injury patient, using pre-transplantation spinal cord function as the control.

DETAILED DESCRIPTION:
The research has carried out in Phase II which is designed as randomized controlled trials.

Selection of patients began in Feb,2013, 48 patients are divided in two group according to a 2:1 ratio (the number of candidates as treated: the candidates as control).

The effectiveness of preliminary trial are evaluated by assessing Frankel/ASIA motor grade, measuring electrophysiological parameters, enhanced MRI and urinary and bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give voluntary (patients may not be able to write) consent.
* Must be able to understand study information provided to him.
* Patients with complete spinal cord < 2 weeks in acute category
* The level of spinal cord injury must be categorized at A level in terms of ASIA Impairment scale.
* Age should be between 19-60 years
* Both male and female

Exclusion Criteria:

* Support respiration by machine
* Melanoma within 5 years
* Infectious diseases including HIV and Hepatitis B, C
* Brain damage or multiple trauma
* Body temperature higher 38 ℃ or acute disorder
* Anemia or thrombocytopenia
* Angina , myocardial infarction , heart disease , embolic disease , chronic renal failure, glomerular disease and chronic obstructive pulmonary disease.
* Congenital or acquired immunodeficiency disorder
* Muscular dystrophy or muscle stiffness
* Non-conscious or voice disorders
* Treatment with cytotoxic drugs ( immunosuppressive drugs , corticosteroids and cytotoxic drugs) during the clinical trials .
* Participating in another clinical trial within 3 months
* Other serious disease or disorder can seriously affect the ability to participate in research.
* Women who are pregnant or lactating .
* Allergy to antibiotics and anesthetics .
* Do not agree to participate in research

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with adverse events after transplantation. | 24 months
  Number of Participants with adverse events is as a measure of safety and tolerability after ADSC transplantation. Adverse events can be impaired liver and kidney, immunosuppression or immune deficiency, hypersensitivity, anaphylactic shock, meningitis symptoms, etc.

SECONDARY OUTCOMES:
Changes of spinal cord edema in the MRI at the lesion site | 24 months
  Patients take MRI at the lesion site before each injection and after transplantation 6 months, 12 months, 24 months. MRI at the lesion site shows spinal cord edema level is reduced or not.
Urinary and bowel function Improvement | 24 months
  Bladder pressure monitory to assess ability to feel and control urination and bowel.
Muscle contraction force measurement | 24 months
  Comparison the electromyography (EMG) score during contraction of given muscles before each injection and after transplantation 6 months, 12 months and 24 months.
Significant clinical improvement in ASIA impairment scale and general condition. | 24 months
  Patients are assess improvement level based on American Spinal Injury Assessment scale of A,B,C,D or E before and after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Phuc Ba Duong, MD, Principal Investigator — Tri Phuoc Biotechnology., JSC; Hoa D Nguyen, MD, Principal Investigator — Vietnamese- German Hospital
Locations (1):
- Vietnamese- German Hospital, Hanoi, Hanoi, Vietnam